CLINICAL TRIAL: NCT06440954
Title: To Investigate the Efficacy and Resistance Mechanisms of Intrathecal Pemetrexed in Advanced Non-small Cell Lung Cancer (NSCLC) Patients Harboring Oncogenic Mutations With Leptomeningeal Metastases
Brief Title: Efficacy and Resistance Mechanisms of IP in NSCLC With Leptomeningeal Metastases
Acronym: EPIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Collaborators: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240442
Record Dates: First submitted 2024-04-23; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrathecal pemetrexed (Experimental): Intrathecal pemetrexed
  Interventions: Drug: Intrathecal pemetrexed

INTERVENTIONS:
Drug: Intrathecal pemetrexed — Intrathecal pemetrexed(50mg) twice a week for 1 week (day 1 and day 5) as induction treatment, then once monthly until progressive disease.
  Other Names: pemetrexed

SUMMARY:
This is a prospective interventional study clinical study to investigate the efficacy and resistance mechanisms of intrathecal pemetrexed in patients with driver gene mutations advanced NSCLC with leptomeningeal metastases.

DETAILED DESCRIPTION:
This is a prospective interventional clinical study aimed at investigating the efficacy and resistance mechanisms of intrathecal pemetrexed in advanced NSCLC patients with EGFR, ALK, and ROS1 mutations presenting leptomeningeal metastases. Approximately 30 advanced NSCLC patients with EGFR, ALK, and ROS1 mutations, who have developed leptomeningeal metastases following TKI resistance, will receive intrathecal pemetrexed. Cerebrospinal fluid samples will be collected before and after pemetrexed resistance to analyze molecular mechanisms and differences. Second-generation gene detection will be performed to identify potential resistance mechanisms to pemetrexed. The study is expected to commence recruitment in mainland China around April 2024, with an anticipated completion date in April 2025.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histopathology or cytology confirmed metastatic non-small cell lung cancer with leptomeningeal metastasis after TKI resistant.
3. EGFR mutant, ALK fusion, ROS1 fusion, and other oncogenic alterations including RET fusion, BRAF mutation, NTRK fusion, KRAS mutation was confirmed by an accredited local laboratory.
4. Adequate bone marrow hematopoiesis and organ function
5. Agree to receive intrathecal pemetrexed
6. ECOG 0 - 2.
7. Predicted survival ≥ 12 weeks.

Exclusion Criteria:

1. Previously received intrathecal pemetrexed therapy for locally advanced or metastatic disease.
2. Subjects who have received any of the following treatments must be excluded:

   Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
3. Presence of spinal cord compression or meningeal metastasis.
4. History of other malignant tumors within 2 years.
5. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
6. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
7. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
8. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
9. Heart-related diseases or abnormalities
10. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
11. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
12. Live vaccine was given 2 weeks before the first medication.
13. Women who are breastfeeding or pregnant.
14. Hypersensitivity to the test drug and the ingredients.
15. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival (I-PFS) | Time from first subject dose to study completion, or up to 36 month
  Intracranial progression-free survival was defined as the duration from the start of IP to the worsening of neurological symptoms, radiological confirmation of brain progression, or patient death

SECONDARY OUTCOMES:
System progression-free survival (s-PFS) | Time from first subject dose to study completion, or up to 36 month
  System progression-free survival was defined as the duration from the start of IP to the worsening of neurological symptoms, radiological confirmation of brain progression, or patient death

OTHER OUTCOMES:
Overall Survival Time | Time from first subject dose to study completion, or up to 36 month
  Overall Survival Time was defined as the duration from the start of IP to patient death

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China